CLINICAL TRIAL: NCT06573138
Title: The Efficacy and Safety of Selinexor, Anti-PD-1 Antibody Plus Golidocitinib in the Treatment of Relapsed or Refractory Natural Killer / T-cell Lymphoma
Brief Title: Selinexor, Anti-PD-1 Antibody Plus Golidocitinib in R/R NKTCL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Prof., Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-NKTCL-4
Record Dates: First submitted 2024-08-16; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Lymphoma, Extranodal NK-T-Cell
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — selinexor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemofree (Experimental): Patients receive 3 cycles of Selinexor, anti-PD-1 antibody plus Golidocitinib.
  Interventions: Drug: Selinexor, anti-PD-1 antibody plus Golidocitinib

INTERVENTIONS:
Drug: Selinexor, anti-PD-1 antibody plus Golidocitinib — Selinexor, 40mg, qw, po; anti-PD1 antibody, 200mg, d1, i.v. (21d cycle); Golidocitinib, Dose 1, 150mg, qod, po; Dose2, 150mg, qd, po.

SUMMARY:
A multicenter, prospective trial to evaluate the efficacy and safety of Selinexor, anti-PD-1 antibody plus Golidocitinib in the treatment of relapsed or refractory Natural Killer / T-cell lymphoma.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy and safety of Selinexor, anti-PD-1 antibody plus Golidocitinib in relapsed or refractory NKTCL and find the optimal treatment regimen for patients with relapsed refractory NKTCL.

Patients receive 3 cycles of Selinexor, anti-PD-1 antibody plus Golidocitinib and then PET evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed histological diagnosis of NKTCL nasal type
2. The subject had received prior adequate anti-lymphoma therapy containing asparaginase
3. Age 14-75 years old
4. expected to live longer than 3 months
5. At least one measurable/evaluable site after diagnostic biopsy before treatment start
6. ECOG performance status of 0-2
7. Adequate hematological and organ function; i.e. ANC >1000 cells /mmc, platelet counts > 50.000/mmc, Hemoglobin > 9 g/dl AST, ALT <3 x ULN; serum bilirubin < 1.5x ULN (patient with Gilbert disease can be enrolled)Serum creatinine < 2 x ULN or creatinine clearance > 50ml/min
8. Tumor tissue (fresh preferred, archival tissue is also acceptable)
9. For women of childbearing potential a negative pregnancy test on day 1 of cycle 1 and agree to adopt adequate measure to avoid pregnancy during study treatment and for at least one year from EOT.
10. For men agreement to remain abstinent or to use barrier contraception
11. Signed Informed consent

Exclusion Criteria:

1. Confirmed histological diagnosis of aggressive NK cell leukemia
2. Evidence of suspect of CNS disease.
3. Has an active autoimmune disease that has required systemic treatment in past 2-years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs), including but not limited to myotonia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associate with antiphospholipid syndrome, wegener's granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis or glomerulonephritis. The following exception are allowed: patients with autoimmune related hypothyroidism or type I diabetes mellitus who are on stable treatment. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
4. Treatment with systemic immunosuppressive medications, including prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide and anti-tumor necrosis factor (anti-TNF) agents within 2 weeks prior to cycle 1 day 1; inhaled corticosteroids are allowed.
5. Active infection requiring systemic therapy
6. History of (non-infectious) pneumonitis that required steroids; evidence of interstitial lung disease or active, non-infectious pneumonitis
7. Significant cardiovascular disease, myocardial infarction in the previous 3 months, unstable arrhythmias, or unstable angina.
8. History of other(s) infiltrating cancer(s) in the previous 3 years that were not treated with curative intent or who are still receiving anticancer therapy (including hormone therapy for breast or prostate cancer).
9. HBsAg, HCV or HIV positivity. Positive serology is admitted for HBV and HCV but DNA/RNA test must be negative
10. Pregnant or lactating women
11. Administration of a live attenuated vaccine within 4 weeks before cyle 1 day 1. Patients must not receive live, attenuate vaccines, including influenza vaccines at any time during study.
12. Other uncontrollable medical condition that may interfere the participation of the study

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Best CRR | through study completion, an average of 1 year
  CRR defined according to 2014 Lugano criteria and 2016 Refinement of the Lugano Classification lymphoma response criteria in the era of immunomodulatory therapy.